CLINICAL TRIAL: NCT04654689
Title: Impact of the Combined Treatment of Curcumin and Resveratrol Liposomed Polyphenols With G04CB02 on the Clinical Improvement of ALS Patients
Brief Title: Impact of the Combined Treatment of Liposomed Polyphenols With G04CB02 on the ALS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Principal Investigator, José Enrique de la Rubia Ortí, Ph, Director, Fundación Universidad Católica de Valencia San Vicente Mártir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UCV/2020-2021/018; 2020-005143-23 (EudraCT Number)
Record Dates: First submitted 2020-11-13; First posted 2020-12-04 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: * Intervention group: 30 patients will be administered daily the combination of Resveratrol (75mg) and Curcumin (200mg) liposomes with G04CB02 (0.5mg), in a single dose for 2 months.
  * Control group: 30 patients, who will receive a placebo with the same dosage pattern and for the same period of time. The placebo will consist of water with sucrose replacing the liposomed polyphenols, and a soft capsule of microcrystalline methylcellulose instead of G04CB02. Both the packaging and the capsule format will be identical to those of the treatment administered in the intervention group.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): 30 patients will be given the combination of resveratrol and curcumin liposomed with G04CB02, in a single daily dose for 2 months.
  Interventions: Dietary Supplement: Liposomed polyphenols resveratrol and curcumin; Dietary Supplement: Isocaloric Diet; Drug: G04CB02
- Control group (Placebo Comparator): 30 patients, who will receive a placebo with the same dosage pattern and for the same period of time. The placebo will consist of water with sucrose replacing the liposomal polyphenols, and a soft capsule of microcrystalline methylcellulose instead of G04CB02. Both the packaging and the capsule format will be identical to those of the treatment administered in the intervention group
  Interventions: Other: Placebo for liposomed resveratrol and curcumin; Dietary Supplement: Isocaloric Diet; Other: Placebo microcrystalline methylcellulose

INTERVENTIONS:
Dietary Supplement: Liposomed polyphenols resveratrol and curcumin — Combination of resveratrol (75mg) and curcumin (200mg) liposomed
  Arms: Intervention group
Other: Placebo for liposomed resveratrol and curcumin — Water with sucrose replacing the liposomed polyphenols
  Arms: Control group
Dietary Supplement: Isocaloric Diet — 40% carbohydrates, 40% lipids and 20% proteins
Drug: G04CB02 — G04CB02, in a single daily dose for 2 months
  Arms: Intervention group
Other: Placebo microcrystalline methylcellulose — Placebo replacing G04CB02
  Arms: Control group

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a disease of an inflammatory nature, which causes progressive muscle weakness associated with cognitive and behavioural disorders. Pathogenically, it is characterised by loss of oxidative control, excitotoxicity due to excess glutamate and intestinal dysbiosis. In the absence of curative treatment, the aim of the study is to assess the impact at a clinical level of the combination of liposomed polyphenols to improve their effectiveness, with the drug G04CB02 which shows great anti-ALS properties by Molecular Topology methodology. A prospective, longitudinal, mixed, analytical, experimental and double-blind study is proposed, with a population sample of 60 patients distributed randomly in 30 patients in the intervention group who will receive treatment for 2 months, and 30 patients in the control group who will receive a placebo for the same period. The assessment will be at time 0, and at 2 months and 4 months after treatment, with functional, cognitive and behavioural tests, and of the state of inflammation and oxidation; and at time 0 and 2 months, of the intestinal microbiota.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is the most common neurodegenerative disease of an inflammatory nature among those affecting motor neurons, with a life expectancy of 3 to 5 years. It is characterised by the loss of motor neurons, and can be of the bulbar type when the pathology begins to affect the motor neurons located in the spinal bulb, or of the medullary type when it begins with a loss of strength and weakness in the extremities. Both types eventually lead to an affectation of both motor neurons that results in progressive paralysis of the voluntary muscles until the patient dies. In addition, the pathology presents cognitive and behavioural alterations. Specifically, deficits have been described in verbal fluency, memory, emotional processing or social cognition, which appear to be mainly associated with hypoperfusion of the prefrontal area or hypometabolism.

Pathogenically, ALS is characterised by an alteration in mitochondrial energy use at a neuronal level, mainly linked to a lower activity of the enzymes of the electron transport chain in the spinal cord. This alteration is a consequence of loss of oxidative control, excessive generation of oxidative free radicals, accumulation of neurofilaments, and excitotoxicity linked to an increase in the neurotransmitter glutamate.

In this respect, it has been suggested that bacterial dysbiosis, related to cognitive and behavioural worsening, could also contribute to this adverse neuroinflammatory state, having been associated with a greater risk of suffering from neurodegenerative diseases. Specifically in ALS, a variation in intestinal microbial composition has recently been observed, with an increased abundance of E. coli and enterobacteria, and a low abundance of total yeast, in patients suffering from ALS; and lower levels of non-butyrate producing bacteria needed to maintain the integrity of the intestinal barrier, immune competition and energy metabolism. In contrast, increased Akkermansia muciniphila has been associated with higher levels of nicotinamide and improved disease symptoms in the animal model of the disease.

This evidence, associated with the lack of medical treatment to cure the disease, makes it necessary to look for new therapeutic alternatives of a non-pharmacological nature. These include the administration of effective antioxidants, which reverse the high oxidative stress and inflammation characteristic of the disease. This type of treatment (specifically the association of the antioxidants Pterostilbene and Nicotinamide riboside) has already been applied by our research group to patients with ALS, achieving significant clinical improvements such as: greater functional capacity, greater respiratory capacity, increased muscle strength and electrical activity in the upper and lower limbs, as well as an increase in the percentage of skeletal muscle associated with fat loss. In this sense, several polyphenols have also been tested in animal models, among which the activity shown by Resveratrol stands out, with a high antioxidant power and great neuroprotective capacity, which is associated with an increase in the expression and activation of SIRT1 and AMPK in the ventral part of the spinal cord after its administration. Both mediators promoted the normalization of autophage flow and, more importantly, increased mitochondrial biogenesis in SOD1-G93A mice. However, their beneficial effects are strongly limited by their low availability. This limitation can be overcome by administering Resveratrol and its natural analogues, incorporated in liposomes or nanoparticles, as this is the best option for guaranteeing stability and bioavailability, after administration and absorption of the antioxidant.

Moreover, the effects of the polyphenol Curcumin have already been studied in ALS. In a paper by Chico et al, its effects were studied in ALS patients at doses of 600mg/day for 6 months. In this study they found that Curcumin generated a slight slowdown in the progression of the disease, improving aerobic metabolism and oxidative damage. Furthermore, the use of nanobiotechnology with Curcumin (80mg/day) in the treatment of ALS patients obtained positive results showing that nanocurcumin is safe and could improve the probability of survival as an additional treatment in these patients, especially those with existing bulbar symptoms. In short, the use of both antioxidants in liposome form improves the bioavailability and effects of both, and their liposome combination has already been successfully tested in vivo in prostate cancer patients.

These anti-ALS effects of the two molecules could be complemented by their action in improving the microbiota. To obtain the bioactive products of Curcumin, biotransformation by the human intestinal microflora is necessary; in a bidirectional manner, it has been demonstrated that Curcumin has beneficial effects on the intestinal microbiota by increasing the number of bacterial families such as: Prevotellaceae, Bifidobacterium, Lactobacilli, Bacteroidaceae and Rikenellaceae, and reducing the number of pro-inflammatory bacterial families such as: Enterobacteria and Enterococci. With regard to Resveratrol, as occurs with Curcumin, the intestinal microflora contributes to its metabolism; and also stands out in the increased production of anti-inflammatory bacteria of the Lactobacillus or Bifidobacterium genera. In addition, it has been found to increase levels of the bacterium Akkermansia Muciniphila, which is associated with an improvement in the prognosis of the disease.

Finally, the use of these two antioxidants in ALS would be combined synergistically by repositioning G04CB02, a drug selected after a molecular topology scan of more than 30,000 drugs from two databases: CMC and Drugbank. It is currently marketed for the treatment of different pathologies, such as benign prostatic hyperplasia and androgenic alopecia. According to the in silico studies based on Molecular Topology carried out by Dr. Gálvez's team, a very promising anti-ALS effect has been identified for G04CB02, linked to the TDP-43 RNA mediator, among others. Drug design using molecular topology consists of applying topological descriptors to identify and describe, using a specific mathematical pattern, molecules and/or drugs related to a specific disease, in this case ALS. Using molecules with proven anti-ALS activity (Edaravone and Riluzole) and the TDP-43 RNA mediator, this mathematical pattern was identified and the databases mentioned above were traced with the aim of identifying drugs that share the same pattern and therefore have potential anti-ALS activity. In addition, considering the current shortage of effective treatments for ALS, other mathematical patterns related to anti-inflammatory, antioxidant, neuroprotective and analgesic activity were taken into account when selecting the G04CB02 candidate. To date, molecular topology has enabled the identification of new treatments for CNS diseases such as Alzheimer's, cancer and very recently SARS-Cov-2, among others.

ELIGIBILITY:
Inclusion Criteria:

* All ALS patients, over 18 years of age and with a clear diagnosis and symptomatology of ALS since at least 6 months.

Exclusion Criteria:

* Women under 50 years of age and childbearing age.
* Tracheotomy patients.
* Patients with invasive or non-invasive ventilation with positive ventilatory pressure
* Patients with evidence of dementia.
* Patients with alcohol or drug abuse dependency.
* Patients infected with B or C hepatitis, or HIV positive
* Renal patients with creatinine levels twice as high as normal markers.
* Liver patients with liver markers (ALT, AST) elevated 3 times above normal levels.
* Patients included in other research with drugs or therapies in the experimental phase.
* Patients treated with anticoagulants or with haemostatic problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
Revised Amyotrophic Lateral Sclerosis Functional Rating Scale associated with ALS | Time 0
  Maximum value: 48 points; Means better outcome motor variables Minimum value: 0 points
Revised Amyotrophic Lateral Sclerosis Functional Rating Scale associated with ALS | 2 months
  Maximum value: 48 points; Means better outcome motor variables Minimum value: 0 points
Revised Amyotrophic Lateral Sclerosis Functional Rating Scale associated with ALS | 4 months
  Maximum value: 48 points; Means better outcome motor variables Minimum value: 0 points
Electromyography | Time 0
  Motor Variables
Electromyography | 2 months
  Motor Variables
Electromyography | 4 months
  Motor Variables
Measurement of forced vital capacity | Time 0
  Motor Variables
Measurement of forced vital capacity | 2 months
  Motor Variables
Measurement of forced vital capacity | 4 months
  Motor Variables

SECONDARY OUTCOMES:
Quantitative measurement of plasma IL-6 and TNF-alpha. | Time 0
  Variables related to inflammation and oxidation
Quantitative measurement of plasma IL-6 and TNF-alpha. | 2 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma IL-6 and TNF-alpha. | 4 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma PCR. | Time 0
  Variables related to inflammation and oxidation
Quantitative measurement of plasma PCR. | 2 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma PCR. | 4 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma haptoglobin. | Time 0
  Variables related to inflammation and oxidation
Quantitative measurement of plasma haptoglobin. | 2 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma haptoglobin. | 4 months
  Variables related to inflammation and oxidation
Quantitative measurement of TEAC (oxidation). | Time 0
  Variables related to inflammation and oxidation
Quantitative measurement of TEAC (oxidation). | 2 months
  Variables related to inflammation and oxidation
Quantitative measurement of TEAC (oxidation). | 4 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma 8-oxoG. | Time 0
  Variables related to inflammation and oxidation
Quantitative measurement of plasma 8-oxoG. | 2 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma 8-oxoG. | 4 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma MDA. | Time 0
  Variables related to inflammation and oxidation
Quantitative measurement of plasma MDA. | 2 months
  Variables related to inflammation and oxidation
Quantitative measurement of plasma MDA. | 4 months
  Variables related to inflammation and oxidation
Edinburgh Cognitive and Behavioral ALS Screen | Time 0
  Variable for cognitive and behavioural assesment
  Maximum value: 136 points; Means better outcome Minimum value: 0 points
  Includes a behavioural test to interview the care provider
Edinburgh Cognitive and Behavioral ALS Screen | 2 months
  Variable for cognitive and behavioural assesment
  Maximum value: 136 points; Means better outcome Minimum value: 0 points
  Includes a behavioural test to interview the care provider
Edinburgh Cognitive and Behavioral ALS Screen | 4 months
  Variable for cognitive and behavioural assesment
  Maximum value: 136 points; Means better outcome Minimum value: 0 points
  Includes a behavioural test to interview the care provider
Frontal Assessment Battery | Time 0
  Variable for cognitive and behavioural assesment
  Maximum value: 18 points; Means better outcome 16-15 points means frontosubcortical deficit 13-12 points means frontosubcortical dementia Minimum value: 0 points
  Includes a behavioural test to interview the care provider
Frontal Assessment Battery | 2 months
  Variable for cognitive and behavioural assesment
  Maximum value: 18 points; Means better outcome 16-15 points means frontosubcortical deficit 13-12 points means frontosubcortical dementia Minimum value: 0 points
  Includes a behavioural test to interview the care provider
Frontal Assessment Battery | 4 months
  Variable for cognitive and behavioural assesment
  Maximum value: 18 points; Means better outcome 16-15 points means frontosubcortical deficit 13-12 points means frontosubcortical dementia Minimum value: 0 points
  Includes a behavioural test to interview the care provider

OTHER OUTCOMES:
Variables related to the microbiota | Time 0
  A Clinical Intestinal Microbiome will be performed, which is an analysis of the bacterial microbiota present in the intestine, from a stool sample.
Variables related to the microbiota | 4 months
  A Clinical Intestinal Microbiome will be performed, which is an analysis of the bacterial microbiota present in the intestine, from a stool sample.

CONTACTS AND LOCATIONS:
Overall Officials: José Enrique De la Rubia Ortí, Ph, Principal Investigator — Catholic University of Valencia
Locations (1):
- José Enrique de la Rubia Ortí, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Variables related to inflammation and oxidation:
  * Quantitative measurement of plasma IL-6 and TNF-alpha.
  * Quantitative measurement of plasma PCR.
  * Quantitative measurement of plasma haptoglobin.
  * Quantitative measurement of TEAC (oxidation).
  * Quantitative measurement of plasma 8-oxoG.
  * Quantitative measurement of plasma MDA.
  Variables for cognitive and behavioural assessment:
  * Edinburgh Cognitive and Behavioral ALS Screen
  * Frontal Assessment Battery (FAB)

REFERENCES:
- [Background] Riancho J, Gonzalo I, Ruiz-Soto M, Berciano J. Why do motor neurons degenerate? Actualization in the pathogenesis of amyotrophic lateral sclerosis. Neurologia (Engl Ed). 2019 Jan-Feb;34(1):27-37. doi: 10.1016/j.nrl.2015.12.001. Epub 2016 Feb 4. English, Spanish. PMID 26853842
- [Background] Gordon PH. Amyotrophic Lateral Sclerosis: An update for 2013 Clinical Features, Pathophysiology, Management and Therapeutic Trials. Aging Dis. 2013 Oct 1;4(5):295-310. doi: 10.14336/AD.2013.0400295. PMID 24124634
- [Background] Woolley SC, Jonathan S Katz. Cognitive and behavioral impairment in amyotrophic lateral sclerosis. Phys Med Rehabil Clin N Am. 2008 Aug;19(3):607-17, xi. doi: 10.1016/j.pmr.2008.04.002. PMID 18625419
- [Background] Phukan J, Pender NP, Hardiman O. Cognitive impairment in amyotrophic lateral sclerosis. Lancet Neurol. 2007 Nov;6(11):994-1003. doi: 10.1016/S1474-4422(07)70265-X. PMID 17945153
- [Background] Ralli M, Lambiase A, Artico M, de Vincentiis M, Greco A. Amyotrophic Lateral Sclerosis: Autoimmune Pathogenic Mechanisms, Clinical Features, and Therapeutic Perspectives. Isr Med Assoc J. 2019 Jul;21(7):438-443. PMID 31507117
- [Background] Ticinesi A, Nouvenne A, Tana C, Prati B, Meschi T. Gut Microbiota and Microbiota-Related Metabolites as Possible Biomarkers of Cognitive Aging. Adv Exp Med Biol. 2019;1178:129-154. doi: 10.1007/978-3-030-25650-0_8. PMID 31493226
- [Background] Alifirova VM, Zhukova NG, Zhukova IA, Mironova YS, Petrov VA, Izhboldina OP, Titova MA, Latypova AV, Nikitina MA, Dorofeeva YB, Saltykova IV, Tyakht AV, Kostryukova ES, Sazonov AE. [Correlation Between Emotional-Affective Disorders and Gut Microbiota Composition in Patients with Parkinson's Disease]. Vestn Ross Akad Med Nauk. 2016;71(6):427-35. doi: 10.15690/vramn734. Russian. PMID 29298003
- [Background] Spielman LJ, Gibson DL, Klegeris A. Unhealthy gut, unhealthy brain: The role of the intestinal microbiota in neurodegenerative diseases. Neurochem Int. 2018 Nov;120:149-163. doi: 10.1016/j.neuint.2018.08.005. Epub 2018 Aug 14. PMID 30114473
- [Background] Roy Sarkar S, Banerjee S. Gut microbiota in neurodegenerative disorders. J Neuroimmunol. 2019 Mar 15;328:98-104. doi: 10.1016/j.jneuroim.2019.01.004. Epub 2019 Jan 9. PMID 30658292
- [Background] Mazzini L, Mogna L, De Marchi F, Amoruso A, Pane M, Aloisio I, Cionci NB, Gaggia F, Lucenti A, Bersano E, Cantello R, Di Gioia D, Mogna G. Potential Role of Gut Microbiota in ALS Pathogenesis and Possible Novel Therapeutic Strategies. J Clin Gastroenterol. 2018 Nov/Dec;52 Suppl 1, Proceedings from the 9th Probiotics, Prebiotics and New Foods, Nutraceuticals and Botanicals for Nutrition & Human and Microbiota Health Meeting, held in Rome, Italy from September 10 to 12, 2017:S68-S70. doi: 10.1097/MCG.0000000000001042. PMID 29782468
- [Background] Wright ML, Fournier C, Houser MC, Tansey M, Glass J, Hertzberg VS. Potential Role of the Gut Microbiome in ALS: A Systematic Review. Biol Res Nurs. 2018 Oct;20(5):513-521. doi: 10.1177/1099800418784202. Epub 2018 Jun 20. PMID 29925252
- [Background] Erber AC, Cetin H, Berry D, Schernhammer ES. The role of gut microbiota, butyrate and proton pump inhibitors in amyotrophic lateral sclerosis: a systematic review. Int J Neurosci. 2020 Jul;130(7):727-735. doi: 10.1080/00207454.2019.1702549. Epub 2019 Dec 23. PMID 31870202
- [Background] Blacher E, Bashiardes S, Shapiro H, Rothschild D, Mor U, Dori-Bachash M, Kleimeyer C, Moresi C, Harnik Y, Zur M, Zabari M, Brik RB, Kviatcovsky D, Zmora N, Cohen Y, Bar N, Levi I, Amar N, Mehlman T, Brandis A, Biton I, Kuperman Y, Tsoory M, Alfahel L, Harmelin A, Schwartz M, Israelson A, Arike L, Johansson MEV, Hansson GC, Gotkine M, Segal E, Elinav E. Potential roles of gut microbiome and metabolites in modulating ALS in mice. Nature. 2019 Aug;572(7770):474-480. doi: 10.1038/s41586-019-1443-5. Epub 2019 Jul 22. PMID 31330533
- [Background] de la Rubia JE, Drehmer E, Platero JL, Benlloch M, Caplliure-Llopis J, Villaron-Casales C, de Bernardo N, AlarcOn J, Fuente C, Carrera S, Sancho D, GarcIa-Pardo P, Pascual R, JuArez M, Cuerda-Ballester M, Forner A, Sancho-Castillo S, Barrios C, Obrador E, Marchio P, Salvador R, Holmes HE, Dellinger RW, Guarente L, Estrela JM. Efficacy and tolerability of EH301 for amyotrophic lateral sclerosis: a randomized, double-blind, placebo-controlled human pilot study. Amyotroph Lateral Scler Frontotemporal Degener. 2019 Feb;20(1-2):115-122. doi: 10.1080/21678421.2018.1536152. Epub 2019 Jan 22. PMID 30668199
- [Background] Song W, Song Y, Kincaid B, Bossy B, Bossy-Wetzel E. Mutant SOD1G93A triggers mitochondrial fragmentation in spinal cord motor neurons: neuroprotection by SIRT3 and PGC-1alpha. Neurobiol Dis. 2013 Mar;51:72-81. doi: 10.1016/j.nbd.2012.07.004. Epub 2012 Jul 20. PMID 22819776
- [Background] Asensi M, Medina I, Ortega A, Carretero J, Bano MC, Obrador E, Estrela JM. Inhibition of cancer growth by resveratrol is related to its low bioavailability. Free Radic Biol Med. 2002 Aug 1;33(3):387-98. doi: 10.1016/s0891-5849(02)00911-5. PMID 12126761
- [Background] Poltronieri P, Xu B, Giovinazzo G. Resveratrol and other Stilbenes: Effects on Dysregulated Gene Expression in Cancers and Novel Delivery Systems. Anticancer Agents Med Chem. 2021;21(5):567-574. doi: 10.2174/1871520620666200705220722. PMID 32628597
- [Background] Chico L, Ienco EC, Bisordi C, Lo Gerfo A, Petrozzi L, Petrucci A, Mancuso M, Siciliano G. Amyotrophic Lateral Sclerosis and Oxidative Stress: A Double-Blind Therapeutic Trial After Curcumin Supplementation. CNS Neurol Disord Drug Targets. 2018;17(10):767-779. doi: 10.2174/1871527317666180720162029. PMID 30033879
- [Background] Ahmadi M, Agah E, Nafissi S, Jaafari MR, Harirchian MH, Sarraf P, Faghihi-Kashani S, Hosseini SJ, Ghoreishi A, Aghamollaii V, Hosseini M, Tafakhori A. Safety and Efficacy of Nanocurcumin as Add-On Therapy to Riluzole in Patients With Amyotrophic Lateral Sclerosis: A Pilot Randomized Clinical Trial. Neurotherapeutics. 2018 Apr;15(2):430-438. doi: 10.1007/s13311-018-0606-7. PMID 29352425
- [Background] Huang M , Liang C , Tan C , Huang S , Ying R , Wang Y , Wang Z , Zhang Y . Liposome co-encapsulation as a strategy for the delivery of curcumin and resveratrol. Food Funct. 2019 Oct 16;10(10):6447-6458. doi: 10.1039/c9fo01338e. PMID 31524893
- [Background] Narayanan NK, Nargi D, Randolph C, Narayanan BA. Liposome encapsulation of curcumin and resveratrol in combination reduces prostate cancer incidence in PTEN knockout mice. Int J Cancer. 2009 Jul 1;125(1):1-8. doi: 10.1002/ijc.24336. PMID 19326431
- [Background] Zam W. Gut Microbiota as a Prospective Therapeutic Target for Curcumin: A Review of Mutual Influence. J Nutr Metab. 2018 Dec 16;2018:1367984. doi: 10.1155/2018/1367984. eCollection 2018. PMID 30647970
- [Background] Luca SV, Macovei I, Bujor A, Miron A, Skalicka-Wozniak K, Aprotosoaie AC, Trifan A. Bioactivity of dietary polyphenols: The role of metabolites. Crit Rev Food Sci Nutr. 2020;60(4):626-659. doi: 10.1080/10408398.2018.1546669. Epub 2019 Jan 7. PMID 30614249
- [Background] Chen ML, Yi L, Zhang Y, Zhou X, Ran L, Yang J, Zhu JD, Zhang QY, Mi MT. Resveratrol Attenuates Trimethylamine-N-Oxide (TMAO)-Induced Atherosclerosis by Regulating TMAO Synthesis and Bile Acid Metabolism via Remodeling of the Gut Microbiota. mBio. 2016 Apr 5;7(2):e02210-15. doi: 10.1128/mBio.02210-15. PMID 27048804
- [Background] Qiao Y, Sun J, Xia S, Tang X, Shi Y, Le G. Effects of resveratrol on gut microbiota and fat storage in a mouse model with high-fat-induced obesity. Food Funct. 2014 Jun;5(6):1241-9. doi: 10.1039/c3fo60630a. Epub 2014 Apr 11. PMID 24722352
- [Background] Sung MM, Byrne NJ, Robertson IM, Kim TT, Samokhvalov V, Levasseur J, Soltys CL, Fung D, Tyreman N, Denou E, Jones KE, Seubert JM, Schertzer JD, Dyck JR. Resveratrol improves exercise performance and skeletal muscle oxidative capacity in heart failure. Am J Physiol Heart Circ Physiol. 2017 Apr 1;312(4):H842-H853. doi: 10.1152/ajpheart.00455.2016. Epub 2017 Feb 3. PMID 28159807
- [Background] Zhao L, Zhang Q, Ma W, Tian F, Shen H, Zhou M. A combination of quercetin and resveratrol reduces obesity in high-fat diet-fed rats by modulation of gut microbiota. Food Funct. 2017 Dec 13;8(12):4644-4656. doi: 10.1039/c7fo01383c. PMID 29152632
- [Background] Slater S, Dumas C, Bubley G. Dutasteride for the treatment of prostate-related conditions. Expert Opin Drug Saf. 2012 Mar;11(2):325-30. doi: 10.1517/14740338.2012.658040. Epub 2012 Feb 8. PMID 22316171
- [Background] Arif T, Dorjay K, Adil M, Sami M. Dutasteride in Androgenetic Alopecia: An Update. Curr Clin Pharmacol. 2017;12(1):31-35. doi: 10.2174/1574884712666170310111125. PMID 28294070
- [Background] Zanni R, Galvez-Llompart M, Garcia-Domenech R, Galvez J. What place does molecular topology have in today's drug discovery? Expert Opin Drug Discov. 2020 Oct;15(10):1133-1144. doi: 10.1080/17460441.2020.1770223. Epub 2020 Jun 4. PMID 32496823
- [Background] Salehi B, Mishra AP, Nigam M, Sener B, Kilic M, Sharifi-Rad M, Fokou PVT, Martins N, Sharifi-Rad J. Resveratrol: A Double-Edged Sword in Health Benefits. Biomedicines. 2018 Sep 9;6(3):91. doi: 10.3390/biomedicines6030091. PMID 30205595
- [Background] Patel KR, Scott E, Brown VA, Gescher AJ, Steward WP, Brown K. Clinical trials of resveratrol. Ann N Y Acad Sci. 2011 Jan;1215:161-9. doi: 10.1111/j.1749-6632.2010.05853.x. PMID 21261655
- [Background] Kuptniratsaikul V, Thanakhumtorn S, Chinswangwatanakul P, Wattanamongkonsil L, Thamlikitkul V. Efficacy and safety of Curcuma domestica extracts in patients with knee osteoarthritis. J Altern Complement Med. 2009 Aug;15(8):891-7. doi: 10.1089/acm.2008.0186. PMID 19678780
- [Background] Deshpande SS, Lalitha VS, Ingle AD, Raste AS, Gadre SG, Maru GB. Subchronic oral toxicity of turmeric and ethanolic turmeric extract in female mice and rats. Toxicol Lett. 1998 May;95(3):183-93. doi: 10.1016/s0378-4274(98)00035-6. PMID 9704820
- [Background] Hewlings SJ, Kalman DS. Curcumin: A Review of Its Effects on Human Health. Foods. 2017 Oct 22;6(10):92. doi: 10.3390/foods6100092. PMID 29065496
- [Background] Chung HT, Noworolski SM, Kurhanewicz J, Weinberg V, Roach Iii M. A pilot study of endorectal magnetic resonance imaging and magnetic resonance spectroscopic imaging changes with dutasteride in patients with low risk prostate cancer. BJU Int. 2011 Oct;108(8 Pt 2):E164-70. doi: 10.1111/j.1464-410X.2010.10061.x. Epub 2011 Mar 24. PMID 21435153
- [Background] Perrotti M, Jain R, Abriel LM, Baroni TE, Corbett AB, Tenenbaum SA. Dutasteride monotherapy in men with serologic relapse following radical therapy for adenocarcinoma of the prostate: a pilot study. Urol Oncol. 2012 Mar-Apr;30(2):133-8. doi: 10.1016/j.urolonc.2010.01.004. Epub 2010 Aug 25. PMID 20800512
- [Background] Kaufmann P, Levy G, Montes J, Buchsbaum R, Barsdorf AI, Battista V, Arbing R, Gordon PH, Mitsumoto H, Levin B, Thompson JL; QALS study group. Excellent inter-rater, intra-rater, and telephone-administered reliability of the ALSFRS-R in a multicenter clinical trial. Amyotroph Lateral Scler. 2007 Feb;8(1):42-6. doi: 10.1080/17482960600888156. PMID 17364435
- [Background] Montes J, Levy G, Albert S, Kaufmann P, Buchsbaum R, Gordon PH, Mitsumoto H. Development and evaluation of a self-administered version of the ALSFRS-R. Neurology. 2006 Oct 10;67(7):1294-6. doi: 10.1212/01.wnl.0000238505.22066.fc. PMID 17030772
- [Background] Witgert M, Salamone AR, Strutt AM, Jawaid A, Massman PJ, Bradshaw M, Mosnik D, Appel SH, Schulz PE. Frontal-lobe mediated behavioral dysfunction in amyotrophic lateral sclerosis. Eur J Neurol. 2010 Jan;17(1):103-10. doi: 10.1111/j.1468-1331.2009.02801.x. Epub 2009 Oct 29. PMID 19874396
- [Background] Butman J, Allegri RF, Harris P, Drake M. [Spanish verbal fluency. Normative data in Argentina]. Medicina (B Aires). 2000;60(5 Pt 1):561-4. Spanish. PMID 11188892
- [Background] Mahone EM, Cirino PT, Cutting LE, Cerrone PM, Hagelthorn KM, Hiemenz JR, Singer HS, Denckla MB. Validity of the behavior rating inventory of executive function in children with ADHD and/or Tourette syndrome. Arch Clin Neuropsychol. 2002 Oct;17(7):643-62. PMID 14591848
- [Background] Portella MJ, Marcos-Bars T, Rami-Gonzalez L, Navarro-Odriozola V, Gasto-Ferrer C, Salamero M. ['Tower of London': mental planning, validity and the ceiling effect]. Rev Neurol. 2003 Aug 1-15;37(3):210-3. Spanish. PMID 12938051
- [Background] Ringholz GM, Appel SH, Bradshaw M, Cooke NA, Mosnik DM, Schulz PE. Prevalence and patterns of cognitive impairment in sporadic ALS. Neurology. 2005 Aug 23;65(4):586-90. doi: 10.1212/01.wnl.0000172911.39167.b6. PMID 16116120
- [Background] Stout JC, Ready RE, Grace J, Malloy PF, Paulsen JS. Factor analysis of the frontal systems behavior scale (FrSBe). Assessment. 2003 Mar;10(1):79-85. doi: 10.1177/1073191102250339. PMID 12675387
- [Background] Galvez, Jorge; Llompart, Javier; Land, David; Pasinetti, Giulio. Compositions for treatment of Alzheimer's disease using AB-reducing and/or AB-anti-aggregation compounds. WO 2010114636 A1 20101636. 2010
- [Background] Galvez, Jorge; Llompart, Javier; Pal, Kollol. N,N-dicyclohexyl-(1S)-isoborneol-10-sulfonamide (MT103) and related compounds for the treatment of cancer. US20040266732. 2004
- [Background] Llompart, Javier; Galvez, Jorge; Pal, Kollol. Treatment of cancer with MT477 derivatives. US20060014770. 2006
- [Background] Gastaminza, P; Garaigorta, U., Benlloch, J.M., Galvez-Llompart, M; Zanni, R, and Galvez, J. Compounds for the treatment and prevention of viral infections caused by coronaviruses. European Patent Application EP20382570.8. 2020
- [Background] Jiménez J, Hernández S, Garcia E, Diaz A, Rodriguez C. Test de atención D2: Datos normativos y desarrollo evolutivo de la atención.Eur J Educ Psychol. 2012; 5: 93-106.
- [Background] Martin R, Hernández S, Rodriguez C, Garcia E. Datos normativos para el Test de Stroop: patrón de desarrollo de la inhibición y formas alternativas para su evaluación. Eur J Educ Psychol. 2012; 5: 39-51
- [Background] Wechsler D. WMS-R: Wechsler Memory Scale-Revised Manual. 1987. San Antonio: The Psychological Corporation
- [Derived] Sancho-Cantus D, Sanchis ES, Casani-Cubel J, Privado J, Escriba J, Carriqui-Suarez AB, Benlloch M, Ceron JJ, Rubio CP, Cubero-Plazas L, de la Rubia Orti JE. Prediction of antioxidant capacity, age, and sex on sleep impairment in patients with amyotrophic lateral sclerosis. Sci Rep. 2025 Jul 1;15(1):21145. doi: 10.1038/s41598-025-07729-5. PMID 40595276
- [Derived] Privado J, Sanchis Sanchis E, Sancho-Cantus D, Cubero-Plazas L, Navarro-Illana E, de la Rubia Orti JE. Prediction of caregiver psychological distress in amyotrophic lateral sclerosis: A cross-sectional study. Rehabil Psychol. 2024 Nov;69(4):364-374. doi: 10.1037/rep0000554. Epub 2024 Jun 20. PMID 38900570